CLINICAL TRIAL: NCT05629026
Title: Study of Lymphatic Dysfunction in Primary and Secondary Lymphedema
Acronym: LYMPHODYS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/22/0128
Record Dates: First submitted 2022-10-03; First posted 2022-11-29 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Intervention Model Description: cross-sectional sample of patients with primary or secondary lymphoedema.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- primary lymphoedema (Experimental): patients with primary lymphoedema
  Interventions: Procedure: Micro-biopsies
- secondary lymphoedema (Experimental): patients with secondary lymphoedema
  Interventions: Procedure: Micro-biopsies

INTERVENTIONS:
Procedure: Micro-biopsies — Two micro-biopsies of limb tissue will be carried out, one on the lymphedema and one in the upper limb not affected.

SUMMARY:
Lymphedema is a disorder of the lymphatic vascular system characterized by impaired lymphatic return and swelling of the extremities and accumulation of undrained interstitial fluid/lymph that results in fibrosis and adipose tissue deposition in the affected area. It can be an inherited condition (primary lymphedema) or occurs after cancer surgery and lymph node removal (secondary lymphedema). It causes a significant morbidity and is a common disabling disease affecting more than 200 million people worldwide, however there is no curative treatment for primary or secondary lymphedema.

DETAILED DESCRIPTION:
Primary lymphedema is an inherited condition whereas secondary lymphedema develops after cancer treatments. Despite common phenotype, a molecular and histological comparison of these two pathologies has never been performed. Primary lymphedema is associated with heterozygous inactivating mutations of the gene encoding vascular endothelial growth factor C and D receptor (VEGFR-3). Primary lymphedema is rare, affecting 1 in 100,000 individuals. Secondary lymphedema is the most common cause of the disease and affects more than 200 million people worldwide.

Secondary lymphedema occurs months, sometimes years after cancer surgery suggesting that lymphedema is not only a side effect of the surgery, but involves modifications of the lymphatic architecture as well as its microenvironment, in particular adipose tissue that accumulates in the limb.

There is no cure for lymphedema because of the lack of identified therapeutic strategies able to restore collecting lymphatic draining function in the arm or in the leg. The goal will be to establish if these pathologies which possess a common denomination exhibit a similar gene expression.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in who developed primary lymphedema or secondary lymphedema after breast cancer treatment.
2. Male and female over the age of 18 and under 75.
3. Patient affiliated to a social security scheme in France.
4. Patient having signed informed consent prior to inclusion in the study and prior to any specific procedure for the study.
5. Patients with no recidive > 3 years after cancer surgery.
6. Patients with Body Mass Index <35.
7. Patient enrolled in a care pathway for the management of their lymphedema (medical and educational care).
8. Patients wearing a compression orthosis on the limb with lymphedema.

Exclusion Criteria:

1. Patients with strong suspicion or with active bacterial or fungal infection.
2. Patient with venous insufficiency associated with lymphedema.
3. Patient with a history of deep venous thrombosis on the limb with lymphedema.
4. History of chronic inflammatory disease.
5. Active neoplasia during parallel management.
6. Patient already included in another therapeutic trial.
7. Pregnant or breastfeeding woman.
8. Metastatic cancer.
9. Bilateral breast cancer.
10. Obliterative arterial disease.
11. Multiple erysipelas.
12. Active smoking (delayed healing).
13. Medicines that may promote delayed healing (Corticosteroid therapy, immunosuppressants).
14. Medication that thins the blood (aspirin and antiplatelet agent, anti-coagulant).
15. Betadine allergy.
16. Patient under guardianship or trusteeship, persons placed under the protection of justice

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of RNA transcripts between lymphoedema limb and healthy limb | Day 1
  The gene expression profile of primary and secondary lymphedema will be determined by high-throughput RNA sequencing (RNAseq) or next-generation sequencing (NGS). It is a molecular methodology that allows the rapid sequencing of thousands to millions of RNA molecules simultaneously, determining the unique and specific order of nucleic acid bases. It is a random sequencing of the whole transcriptome which is used to identify and quantify the RNA resulting from the transcription of the genome at a given time.

SECONDARY OUTCOMES:
LYVE-1 expression in primary and secondary lymphedema by immuno-histology | Day 1
  LYVE-1 (lymphatic vessel endothelial hyaluronan receptor-1) will be determined from immunodetection and staining performed on paraffin sections of lymphedema tissue in comparison with healthy tissue
Podoplanin expression in primary and secondary lymphedema by immuno-histology | Day 1
  Podoplanin expression will be determined from immunodetection and staining performed on paraffin sections of lymphedema tissue in comparison with healthy tissue
Chromatography analysis of Lipids in adipose tissues from primary and secondary lymphoedema | Day 1
  To describe lipid profile in adipose tissues from primary and secondary lymphoedema, in comparison to the healthy limb by chromatography analysis expressed in pg lipid/mg protein.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Malloizel-Delaunay, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No